CLINICAL TRIAL: NCT02375412
Title: Preoperative Evaluation of Autonomic Nervous System by Heart Rate Variability as a Predictor of Postoperative Outcome in the Patient Undergoing Major Elective Abdominal Surgery
Brief Title: Preoperative Measurement of Heart Rate Variability as a Predictor of Postoperative Outcome
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-KARIM-2
Record Dates: First submitted 2015-02-24; First posted 2015-03-02 (Estimated); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: Major Abdominal Surgery
Keywords: heart rate variability; post-operative outcome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pre-operative HRV group: Pre-operative measurement of heart rate variability in patients undergoing elective major abdominal surgery.
  Interventions: Procedure: Pre-operative measurement of heart rate variability

INTERVENTIONS:
Procedure: Pre-operative measurement of heart rate variability — Pre-operative measurement of heart rate variability in patients undergoing elective major abdominal surgery

SUMMARY:
The purpose of the study is to confirm the hypothesis that a dysfunction of the autonomic nervous system could complicate the postoperative course in the patient undergoing surgery. Measurement of heart rate variability (HRV) is a non-invasive method for evaluation of the autonomic nervous system.

DETAILED DESCRIPTION:
The autonomic nervous system (ANS) plays an important role in the maintenance of systemic homeostasis. The homeostasis is modified continually by internal and external stimuli to which the autonomic nervous system modulates the response of organism by tight control on essential functions such as circulation, respiration, hormonal secretion and thermoregulation. Dysfunction of the autonomic nervous system could complicate the perioperative course in the patient undergoing surgery; therefore it should be considered as another risk factor during preoperative evaluation. Nowadays the evaluation of the autonomic nervous system function like a tool for prediction postoperative outcome is not considered in daily anaesthesiology practice. Measurement of heart rate variability (HRV) is a method for evaluation the autonomic nervous system function. It is a non-invasive method that provides information about the autonomic regulation of organism and thus it identifies patients with the autonomic nervous system dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and above
* anticipated duration of surgery more than 120 minutes
* estimated blood loss exceeding more than 15% of blood volume
* American Society of Anesthesiology (ASA) classification 2 or 3

Exclusion Criteria:

* pregnant or lactating women
* age below 21 years of age
* emergency surgery
* American Society of Anesthesiology (ASA) classification 1
* sepsis and septic shock
* severe cardiac arrhythmias

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective major abdominal surgery.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Actual)
Dates: Start 2015-02; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Pre-defined postoperative complications for up to 28 days after surgery | 24 months
  The followed postoperative complications include infectious, respiratory, cardiovascular, abdominal, renal complications, massive postoperative bleeding and preoperative death.

SECONDARY OUTCOMES:
The length of hospitalization | 24 months
  Length of hospital stay will be obtained from the patient record.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Ostrava, Ostrava-Poruba, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laitio T, Jalonen J, Kuusela T, Scheinin H. The role of heart rate variability in risk stratification for adverse postoperative cardiac events. Anesth Analg. 2007 Dec;105(6):1548-60. doi: 10.1213/01.ane.0000287654.49358.3a. PMID 18042846
- [Background] Mazzeo AT, La Monaca E, Di Leo R, Vita G, Santamaria LB. Heart rate variability: a diagnostic and prognostic tool in anesthesia and intensive care. Acta Anaesthesiol Scand. 2011 Aug;55(7):797-811. doi: 10.1111/j.1399-6576.2011.02466.x. Epub 2011 Jun 9. PMID 21658013
- [Background] Heart rate variability. Standards of measurement, physiological interpretation, and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Eur Heart J. 1996 Mar;17(3):354-81. No abstract available. PMID 8737210